CLINICAL TRIAL: NCT00016185
Title: Phase I Study Of Flavopiridol And Docetaxel (Taxotere) In Patients With Advanced Cancers
Brief Title: Flavopiridol and Docetaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068605; P30CA022453 (NIH); WSU-C-2197; NCI-1610
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — alvocidib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: alvocidib
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining flavopiridol and docetaxel in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxic effects and maximum tolerated dose of flavopiridol and docetaxel in patients with advanced solid tumors.
* Determine the objective response rate and duration of response in patients treated with this regimen.
* Determine the pharmacokinetics of these drugs in this patient population.

OUTLINE: This is a dose-escalation study.

Patients receive docetaxel IV over 60 minutes on day 1 and flavopiridol IV continuously over 24 hours on day 2. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel and flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study within 9-11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or unresectable solid tumor

  * No standard relatively effective curative or palliative measures exist
* Measurable disease in at least 1 dimension

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No known clinically active and uncontrolled brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2
* Karnofsky 60-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* ALT/AST no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine normal

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No prior allergic reactions to compounds of similar chemical or biologic composition to flavopiridol or docetaxel
* No other uncontrolled concurrent illness that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situations that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* At least 6 months since prior taxane therapy
* At least 4 weeks since other prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except contraceptives, appetite stimulants, or replacement steroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2003-02 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] El-Rayes BF, Gadgeel S, Parchment R, Lorusso P, Philip PA. A phase I study of flavopiridol and docetaxel. Invest New Drugs. 2006 Jul;24(4):305-10. doi: 10.1007/s10637-005-4343-5. PMID 16683073
- [Result] Patel B, El-Rayes BF, Gadgeel SM, et al.: A phase I study of flavopiridol and docetaxel. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-932, 2003.